## Musically-Guided Paced Breathing Improves Mental Health in War-Affected

## Adolescents

NCI Number: NCT06988800

Consent Form (English)

January 21, 2024



Dear parent/guardian of the esteemed student, After Greetings

DESCRIPTION: A study will be carried out on a sample of high school students from the ninth, tenth, eleventh, and twelfth grades with the aim of reducing anxiety and increasing resilience. Student participants in the study will be asked to answer some questions about their wellbeing, watch videos or participate in other activities and answer questions about their experience of those videos/activities during and after the study is finished. Data on the participant's demographics, thoughts, and feelings will be securely stored. Any identifying information will be removed from the data before sharing with our research partner, Muvik Labs, for analysis and evaluation purposes to improve your experience.

TIME INVOLVEMENT: Student participation will take approximately 10 minutes per day, 2 days a week for up to 12 weeks (not including scheduled breaks at the study site). Participants will also be asked to complete questionnaires about their thoughts and feelings multiple times throughout the study. Before the program begins, at designated times during the study, at the end of the study period, and approximately three months after the end of the program. At each session, questionnaire completion should take approximately 30 minutes.

RISKS AND BENEFITS: Every measure will be taken to secure all confidential data including how it is collected and stored. The benefits which may reasonably be expected to result from this study are improved engagement in classes and a reduction in stress and/or anxiety. We cannot guarantee that students will receive any benefits from this study. Your child's decision whether or not to participate in this study will not affect their grades, treatment, or any other aspect of their engagement in school.

Identifiers will be removed from identifiable private information and, after such removal, the information could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you.

PAYMENTS: Students will receive no payment for their participation. There will also be no cost for participation.

PARTICIPANT'S RIGHTS: The individual privacy of participants will be maintained in all published and written data resulting from the study. If you and your child have read this form and have decided to participate in this study, please understand your child's participation is voluntary and you have the right to withdraw consent or discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled. The only alternative is not to participate. Students have the right to refuse to answer particular questions. The results of this research study may be presented at scientific or professional meetings or published in scientific journals.

Meetings may be held outside normal office or school hours as a part of this study.

| For parents |
|--------------------------------------------------------------------|
| After greetings and appreciation |
| I received your letter, and I allow my son/daughter to participate |
| The student's father/s/ |
| Identification Number / |
| Mobile / Telephone / |



Signature / .....